CLINICAL TRIAL: NCT06747481
Title: Neutrophil-to-lymphocyte Ratio and CA 19.9 as Predictors of Perineural Invasion in Pancreatic Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Pau Plá Sánchez, Medical Doctor, Clinical Investigator, University of Las Palmas de Gran Canaria
Other Study IDs: 2024-260-1
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Cancer, Adult; Perineural Invasion; Neutrophil-to-Lymphocyte Ratio; CA 19.9
Keywords: pancreatic cancer; perineural invasion; Neutrophil-to-Lymphocyte Ratio; CA 19.9
MeSH Terms: conditions — Pancreatic cancer, adult; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pancreatic cancer has an incidence of 1,401,450 new cases diagnosed annually worldwide and is the third leading cause of cancer-related death in Spain. This disease is associated with a poor prognosis, reflected by a 5-year survival rate of less than 5% when all stages are grouped together.

Several prognostic factors for pancreatic cancer have been identified. The most relevant include preoperative levels of carbohydrate antigen 19-9 (CA 19.9), surgical margins after resection, venous and/or arterial vascular involvement, and histopathological features such as affected locoregional lymph nodes, or perineural and lymphovascular invasion. Among all these factors, perineural invasion may be the primary independent factor affecting prognosis, particularly in patients with relatively favorable pathological features.

The identification of perineural invasion before surgery could influence the clinical management of these patients. It may facilitate risk stratification, allowing the identification of patients who would benefit most from neoadjuvant treatments or more aggressive surgical procedures, such as vascular resections. However, perineural involvement is very difficult to detect preoperatively.

Only a few studies have analyzed the possible relationship between CA 19.9 and perineural invasion, and their results are inconsistent. Alternatively, some studies have demonstrated the utility of preoperative multidetector computed tomography in detecting extrapancreatic perineural invasion. However, these radiological tests are still not useful for directly detecting microscopic perineural invasion, especially in early stages.

On the other hand, in recent years, evidence has supported that the systemic inflammatory response may play an important role in the prognosis of different malignancies. Among these inflammatory markers, the neutrophil-to-lymphocyte ratio (NLR) has gained prominence. Regarding pancreatic cancer, many studies suggest that elevated preoperative NLR levels are associated with a worse prognosis. However, no studies have yet been published analyzing a possible relationship between this inflammatory marker and perineural invasion.

The main objective of this study is to correlate the neutrophil-to-lymphocyte ratio (NLR) and CA 19.9 with histopathologically confirmed perineural invasion and, in this way, investigate these data as potential preoperative markers of perineural invasion in pancreatic cancer. Our working hypothesis is that preoperative NLR and CA 19.9 are potential markers of perineural invasion.

As secondary objectives, we aim to study the effect of neoadjuvant therapy on inflammatory markers (NLR) and tumor markers (CEA and CA 19.9) in pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a histopathological diagnosis of adenocarcinoma.
* Surgical resection of the neoplasm.
* Preoperative blood count allowing calculation of the neutrophil-to-lymphocyte ratio and preoperative CA 19.9, both before and after neoadjuvant therapy.

Exclusion Criteria:

* Patients with a diagnosis of another histological type.
* Patients with incomplete data.
* Patients who were not operated on.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with pancreatic cancer and operated on between January 2020 and December 2024 from the participating centers who meet all the inclusion criteria and none of the exclusion criteria will be included.
Sampling Method: Non-Probability Sample
Enrollment: 323 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Perineural invasion | Within 30 days prior to surgery (for NLR and CA 19.9) and immediately following surgery for histopathological confirmation
  The correlation between the preoperative neutrophil-to-lymphocyte ratio (NLR) and CA 19.9 with the presence of histopathologically confirmed perineural invasion in patients with pancreatic cancer

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria, Las Palmas, Spain